CLINICAL TRIAL: NCT04163172
Title: Elbow Hemiarthroplasty Versus Open Reduction and Internal Fixation for AO/OTA Type C2 and C3 Fractures of Distal Humerus in Patients Aged 50 Years or Above; a Randomized Controlled Trial
Brief Title: Elbow Hemiarthroplasty Versus ORIF for Distal Humeral Fractures
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Herlev and Gentofte Hospital (Other)
Responsible Party: Principal Investigator, Ali Al-Hamdani, Medical doctor, shoulder and elbow surgeon., Herlev and Gentofte Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EVORI
Record Dates: First submitted 2019-10-31; First posted 2019-11-14 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Distal Humerus Fracture; Comminuted Fracture; Intra-Articular Fractures
MeSH Terms: conditions — Humeral Fractures, Distal; Fractures, Comminuted; Intra-Articular Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Elbow hemiarthroplasty (Active Comparator): The Latitude anatomical hemiarthroplasty (WRIGHT -Memphis, Tennessee) for distal humeral fractures.
  Interventions: Procedure: Surgical treatment of distal humeral fracture with elbow hemiarthroplasty
- Open reduction and internal fixation (Active Comparator): Double plating (Synthes - Switzerland and West Chester, Pennsylvania, United States) for distal humeral fractures.
  Interventions: Procedure: Surgical treatment of distal humeral fracture with double plating.

INTERVENTIONS:
Procedure: Surgical treatment of distal humeral fracture with elbow hemiarthroplasty — Latitude anatomical elbow hemiarthroplasty (WRIGHT -Memphis, Tennessee)
  Arms: Elbow hemiarthroplasty
Procedure: Surgical treatment of distal humeral fracture with double plating. — Double plating (Synthes - Switzerland and West Chester, Pennsylvania, United States)
  Arms: Open reduction and internal fixation

SUMMARY:
This is a randomized control trial comparing the outcome of ORIF (open reduction and internal fixation) with EHA (elbow hemiarthroplasty) for distal humeral fractures in patients aged 50 years or above.

DETAILED DESCRIPTION:
Intraarticular distal humeral fractures AO/OTA type C2 and C3 pose a surgical challenge despite the evolution of surgical implants and techniques. Open reduction and internal fixation (ORIF) is often preferred as the first choice of treatment, but the results are varying, and sometimes disappointing. Total elbow arthroplasty (TEA) has been widely used for fractures that are not amenable to ORIF in elderly patients, but the mechanical complications remain a challenge, especially in active patients. Elbow hemiarthroplasty (EHA) provides a modern alternative that might avoid the mechanical complications and weight bearing restrictions related to the linked articulation in semiconstrained TEA. There are no studies comparing the results of EHA to that of TEA or ORIF, but case series have reported promising results.

In this study, forty-four patients with AO/OTA type C2 or C3 fractures of distal humerus will be randomized to either ORIF or EHA. The patients will be examined after the operation and at 3 months and 1, 2, 5 and 10 years after the surgery. The main objective of this study is to investigate the best treatment option for distal humeral fractures in patients aged 50 years or above. This can be of value to future patients sustaining these complicated fractures.

ELIGIBILITY:
Inclusion Criteria:

1. Distal humeral fracture AO/OTA type C2 or C3 confirmed by plain radiographs with 2 perpendicular views and CT scan.
2. ASA score 1-3 and physically fit for surgery.
3. Age of 50 years or above.

Exclusion Criteria:

1. Patients unable to follow the rehabilitation protocol or answer the Danish questionnaires because of physical or cognitive inabilities as evaluated by the recruiting surgeon.
2. Significant elbow osteoarthritis as evaluated by the recruiting surgeon based on plain radiographs and CT scan.
3. Fractures that are older than 6 weeks.
4. Other associated elbow fractures.
5. Pathological fractures or relevant elbow pathology.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Oxford Elbow Score (OES) | 2 years after surgery.
  The OES is a 12-item patient-administrated questionnaire that measures the quality of life in patients with elbow disorder. There are three unidimensional domains: Elbow function, pain, and social-psychological status. Each question is answered on a 5-point scale with each question contributing equally to the total score.Thus, the total score ranges from 12-60, with 60 being the worst. For ease of presentation the score is converted to a scale from 0-48 with 48 being the best. The outcome can be interpreted based on a 48-point scale: 0 - 19 - poor; 20-29 - fair; 30-39 - good; and 40-48 - excellent. The Danish version which will be used in this study, has been translated and cultural adapted according to the guidelines by Guillemin, Bombardier and Beaton.

SECONDARY OUTCOMES:
Mayo Elbow Performance Score (MEPS) | 3 months after surgery and 1, 2, 5, and 10 years after surgery.
  The MEPS is a surgeon-administrated instrument that evaluates the outcome after elbow surgery. There are four domains including: Pain (0-45 points), range of motion (0-20 points), stability (0-10 points) and difficulties in daily activities (0-25 points).The outcome can be interpreted based on a 100 points scale: 0 - 60 - poor; 60-74 - fair; 75-89 - good; and 90-100 - excellent.
Pain severity score (VAS) | 3 months after surgery and 1, 2, 5, and 10 years after surgery.
  Pain is answered on a visual analogue scale (VAS) ranging from 0 to 10, with 10 being the worst and 0 represents a pain free elbow.
Range of motion | 3 months after surgery and 1, 2, 5, and 10 years after surgery.
  Measuring the flexion/extension and supination/pronation arcs in degrees.
Patients satisfaction | 3 months after surgery and 1, 2, 5, and 10 years after surgery.
  Patients satisfaction of the treatment will be recorded using 5-items score with 1 being the worst and 5 represents a very satisfied patient.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Al-Hamdani, MD, Principal Investigator — Herlev and Gentofte University Hospital
Locations (1):
- Herlev and Gentofte University Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Al-Hamdani A, Rasmussen JV, Holtz K, Olsen BS. Elbow hemiarthroplasty versus open reduction and internal fixation for AO/OTA type 13 C2 and C3 fractures of distal humerus in patients aged 50 years or above: a randomized controlled trial. Trials. 2020 Jun 8;21(1):497. doi: 10.1186/s13063-020-04418-8. PMID 32513252